CLINICAL TRIAL: NCT03444610
Title: Can we Transfuse Blood Over Shorter Period ?
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase 1 studies are not performed in Saudi Arabia yet
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB 2017-63
Record Dates: First submitted 2018-02-13; First posted 2018-02-23 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Blood Transfusion Complication
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm (blood transfusion escalation rate) (Other): The intervention for the arm (blood transfusion escalation rate) will be about giving blood transfusion with escalating rate as described in intervention part to Any condition that expected to receive more than one blood transfusion, like thalassemia major or intermedia, sickle cell anemia, aplastic anemia, malignant diseases.
  Interventions: Biological: Blood transfusion escalation rate

INTERVENTIONS:
Biological: Blood transfusion escalation rate — 3+3 dose escalation (3 patients/cohort) each started on a fixed rate (standard is 5 ml/kg/ hr).1st cohort start at 6ml/kg/hr till complete prescribed volume. Rate escalation by 1ml/kg/each cohort until dose limiting toxicities (DLTs) or max of 10ml/kg/hr. If no DLTs new cohort enrolled at the next planned rate. If DLTs seen in 1 patient in the cohort, another 3 patients treated with the same dose level.1ry phase I end point is maximum-tolerated rate (MTR) of blood transfusion that can be infused safely ( max rate at which 1 or fewer of 3 patients experienced DLT) or dose of 10ml/kg/hr. DLT is transfusion related adverse event lead to stop of transfusion. MTR is highest dose at which no more than 1of 6 patients experienced a DLT.15 additional patients enrolled at MTR to confirm safety.

SUMMARY:
Blood transfusion is very lengthy procedure and consumes a substantial time from patients and health care providers. On average, it may take most if not all the working day which leads to significant constrains on hospital bed utilization. It starts from pre-transfusion testing, clinical assessment, actual administration of blood and post-transfusion care. The main bulk of this procedure is usually related to administration of the blood which typically given over 3 hours (5ml/kg/hour), although there is no strong evidence to support that. Indeed, it has been accepted as standard of care to transfuse blood over short time as in emergency situations.

OBJECTIVE:

To determine the maximum tolerated blood transfusion rate that can be safely delivered in patient who required blood transfusion i.e. transfusing blood over short time.

METHOD:

This is a phase I, open label, nonrandomized, prospective and rate-finding study. A well-known dose escalation design called 3+3 design will be used to identify the maximum tolerated rate. To assure the safety of such procedure, blood transfusion rate will be escalated very slowly by 1 ml/kg/hour for each cohort until rate-limiting toxicities or maximum of 10ml/kg/hour.

DETAILED DESCRIPTION:
Blood transfusion is the mainstay of care for patients with different types of chronic severe anemia like thalassemia major. However, it is associated with serious risks and complications. In addition, blood transfusion is a lengthy procedure starting from pre-transfusion testing, clinical assessment, actual administration of blood and post-transfusion care. The main bulk of this procedure is usually related to administration of the blood which typically given over 3 hours (5ml/kg/hour) or even longer in certain cases. On average, such procedure may take most if not all the working day which leads to significant constrains on hospital bed utilization. Also, it is a significant burden on the patient and his/her family to comply with chronic transfusion program. As consequences, this leads to repeated absences from work or school.

Although, it is the standard of care to infuse blood at rate of 5ml/kg/hour, there is no strong evidence to support that especially in pediatric population. Indeed, it has been accepted as standard of care to transfuse blood over short time in certain cases. For instance, in an emergency situation, it is allowable to infuse blood over less than one hour. Infusion of stem cells is allowed to be given over one hour as well without a major adverse event. In addition, blood donation is usually done over 30 - 60 minutes. As such, the goal for conducting this study is to find out if we can transfuse blood over the short time without causing any harm.

Transfusion associated circulatory overload (TACO) is one of the complications of blood transfusion and known to occur more in adult patients with specific risk factors. TACO is very rare phenomenon in pediatric patients with normal underlying cardiorespiratory functions. In Literature review in pediatrics there was only one case report and that patient had a significant other co-morbidities and risk factors.

In our study, there will be many safety measures taking in our consideration starting by very selective criteria to roll the patients in the study with clear inclusion and exclusion points. Blood transfusion rate determine during the study and will be escalated by 1ml/kg per each cohort only and before starting the blood transfusion vital signs will be taken then 15 minutes after blood transfusion running and by the end of the procedure so there will be 3 times documented vital signs and for more safety issue the patients will be attached to cardiopulmonary monitoring during the whole procedure. Our patients will have ECHO pre-and post-transfusion to detect right ventricle load. Patients will have Brain natriuretic peptide (BNP) level will be done before and after finishing of blood transfusion.

Then at the end, 24 hours post transfusion evaluation will be done for all patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* Any condition that expected to receive more than one blood transfusion, like thalassemia major or intermedia, sickle cell anemia, aplastic anemia, malignant diseases.
* Age range of 3.0-14 years, inclusive, at the time of study entry.
* Parent or guardian willing and able to provide informed consent.
* Ability to comply with study-related treatments, evaluations, and follow-up.
* Normal Echo study that had been done in the last year.

Exclusion Criteria:

* Inability to receive or tolerate chronic red blood cell (RBC) transfusion therapy, due to any of the following:
* Multiple RBC alloantibodies making cross-matching difficult or impossible.
* RBC autoantibodies making cross-matching difficult or impossible.
* Life threatening condition like shock.
* Hemodynamically unstable.
* Hypoxia with oxygen saturation less than 92% on room air.
* Any patient with signs of respiratory distress (using accessory muscle or acting ala nasi).
* Fluid balance more than 1 liter.
* Known severe allergy (anaphylaxis) to blood transfusion.
* Previous history of Transfusion associated circulatory overload (TACO).
* Heart failure or poor ejection fraction less than 60%.
* Current use of therapeutic agents for heart failure or arrhythmia.
* Newly diagnosed with active cancers in the 1st week of induction therapy.
* Severe anemia- Hb <6gm/dl at the day of transfusion.
* Serum creatinine more than twice the upper limit for age.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-05-31 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
can we transfuse blood over shorter period? | 1 year
  primary out come is transfusion associated circulatory overload(TACO), The Frequency will be used in the study to measure the primary outcome (TACO).